CLINICAL TRIAL: NCT07236775
Title: Evaluation of the Apical Root Resorption in Young Adults Caused by Orthodontic Treatment of Class I Severe Crowding Cases Using Clear Aligners Versus Traditional Fixed Appliances: A Randomized Controlled Clinical Trial
Brief Title: Treatment Outcome of Clear Aligner and Traditional Fixed Appliances in Four Premolar Extraction Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-6-2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Malocclusion, Class I/II; Crowding, Tooth
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clear Aligners (Experimental): Patients in this group will be treated using clear aligners.
  Interventions: Device: Clear Aligners
- Fixed appliances (Active Comparator): Patients in this group will be treated using ordinary fixed appliances.
  Interventions: Device: Traditional fixed appliances

INTERVENTIONS:
Device: Clear Aligners — In-house 3D-fabricated clear aligners will be used.
  Arms: Clear Aligners
Device: Traditional fixed appliances — The ordinary metallic braces will be used in a conventional manner.
  Arms: Fixed appliances

SUMMARY:
Patients with severe crowding requiring the extraction of four premolars will be enrolled in this study. The degree of apical root resorption associated with using the clear aligner technique compared with vestibular fixed appliances in the treatment of severe crowding malocclusion cases requiring the extraction of first premolars will be evaluated using cone beam computed tomography (CBCT) volumes.

There are two groups:

First group (Experimental): the patients in this group will be treated using clear aligners.

Second group (Control): the patients in this group will be treated using fixed appliances.

DETAILED DESCRIPTION:
With the increasing number of young adults requesting esthetic orthodontic treatment, clear aligners have continued to gain widespread use, driven by greater consideration of esthetic aspects and oral health-related quality of life compared to traditional fixed orthodontic appliances. Recently, clear aligners have been used in more complex malocclusion cases that require premolar extraction. Teeth root resorption occurs due to physiological or pathological causes that lead to loss of tooth structure. Apical root resorption (ARR) is a common side effect of orthodontic treatment that requires careful investigation of its location and frequency.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-25 years.
* Class I malocclusion with severe dental crowding.
* Tooth size-arch discrepancy more than 6 mm.
* No congenitally missing or extracted teeth (except for the wisdom teeth).
* No history of previous trauma to the maxillofacial region or surgical interventions.

Exclusion Criteria:

* Previous orthodontic treatment.
* Presence of previously occurred ARR.
* Patients with psychological abnormalities or systemic diseases.
* Patients with known allergies to latex or plastic materials.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Change in root length | First assessment: one day before the commencement of treatment (i.e., initiating orthodontic tooth movement). Second assessment: one day following the end of treatment (which is expected to occur within 12 to 18 months).
  The maximum linear lengths between the root apex and incisal edges (for the anterior teeth) or the cusp tips (for the posterior teeth) will be measured on the cone-beam computed tomography (CBCT) images.
  Differences between the measurements of each tooth before and after treatment provided the amount of apical root resorption in mm.
  The variable will be measured for each tooth (from the central incisors to the first molars) and on both jaws.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Younis Hajeer, Study Director — Faculty of Dentistry, University of Damascus; Samer T. Jaber, Principal Investigator — Faculty of Dentistry, University of Damascus
Locations (1):
- Department of Orthodontics, Faculty of Dentistry, University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaber ST, Hajeer MY, Burhan AS, Alam MK, Al-Ibrahim HM. Treatment effectiveness of young adults using clear aligners versus buccal fixed appliances in class I malocclusion with first premolar extraction using the ABO-Objective Grading System: A randomized controlled clinical trial. Int Orthod. 2023 Dec;21(4):100817. doi: 10.1016/j.ortho.2023.100817. Epub 2023 Oct 12. PMID 37837842
- [Background] Jaber ST, Hajeer MY, Sultan K. Treatment Effectiveness of Clear Aligners in Correcting Complicated and Severe Malocclusion Cases Compared to Fixed Orthodontic Appliances: A Systematic Review. Cureus. 2023 Apr 29;15(4):e38311. doi: 10.7759/cureus.38311. eCollection 2023 Apr. PMID 37128600
- [Background] Jaber ST, Hajeer MY, Burhan AS. The Effectiveness of In-house Clear Aligners and Traditional Fixed Appliances in Achieving Good Occlusion in Complex Orthodontic Cases: A Randomized Control Clinical Trial. Cureus. 2022 Oct 10;14(10):e30147. doi: 10.7759/cureus.30147. eCollection 2022 Oct. PMID 36246088
- [Background] Jaber ST, Hajeer MY, Burhan AS, Latifeh Y. The Effect of Treatment With Clear Aligners Versus Fixed Appliances on Oral Health-Related Quality of Life in Patients With Severe Crowding: A One-Year Follow-Up Randomized Controlled Clinical Trial. Cureus. 2022 May 30;14(5):e25472. doi: 10.7759/cureus.25472. eCollection 2022 May. PMID 35663697